CLINICAL TRIAL: NCT01436344
Title: Markers of Paroxysmal Atrial Fibrillation in Esophageal Holter Electrocardiography
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Commission for Technology and Innovation (Other)
Responsible Party: Rolf Vogel, MD, MD-PhD, University Hospital Bern, Dept. of Cardiology
Other Study IDs: 084/11
Record Dates: First submitted 2011-09-12; First posted 2011-09-19 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation; Atrial Premature Complexes
Keywords: esophageal electrocardiography; electrocardiography; atrial electrogram; atrial function, left
MeSH Terms: conditions — Atrial Fibrillation; Atrial Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Cases: 30 patients with known paroxysmal atrial fibrillation (pAF) will consecutively be recruited from the cardiology ward and the cardiological ambulatory. They will form the "cases" group.
- 2: Controls: For every case patient, an age (+/- one year) and gender matched control person (n=30) without known paroxysmal atrial fibrillation will be included and matched to every case patient.

SUMMARY:
With the use of esophageal Holter electrocardiography (eECG), the investigators will look for surrogate markers of paroxysmal atrial fibrillation. To do so, the investigators will record eECGs in patients with known paroxysmal atrial fibrillation but at the time of eECG-recording in sinus rhythm. To identify markers, the eECGs of those patients will be compared to a group of controls in sinus rhythm without atrial fibrillation. The investigators hypothesis is that it is possible to identify surrogate markers in patients with paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Background

The fast and correct diagnosis of heart rhythm disorders is very important to reduce morbidity and mortality in cardiovascular patients. Atrial fibrillation is of special interest, because it is an important cause of devastating brain strokes. A significant number of strokes has a cardioembolic genesis due to paroxysmal atrial fibrillation which was not diagnosed early enough. Therefore, it is very important to detect atrial fibrillation as soon as possible. With oral anticoagulation an effective therapeutic option in available to prevent cardioembolisms.

In the clinical routine, mostly 24-hour or 7-day ECGs are made to look for cardiac arrhythmias. The use uf such devices is well established. Nevertheless, they have some side effects/limitations. Skin electrodes used for derivation of the ECG often cause skin irritation, sometimes leading to premature termination of the recording. Because of dryout of the contact gel (causes artifacts), small p-waves and especially also motion artifacts, triggered recording or semi-automatic analysis of the recording is problematic, but for longer recording times such a semi-automatic analysis would be helpful. As an alternative esophageal electrocardiography can be performed. Signal quality of the ECG recording (especially of the left atrium) is better than in the standard surface ECG because of the vicinity of the esophagus and the left atrium. The esophagus tolerates well foreign bodies as we know from long-term nasogastric intubation. Therefore use of the esophageal technique for long-term rhythm monitoring is an interesting and promising alternative to conventional surface Holter ECGs.

The diagnosis of paroxysmal atrial fibrillation (pAF) can only be made if an episode of atrial fibrillation occurs during the long-term ECG recording. Surrogate markers of pAF could identify a "population at risk" in which pAF has to be suspected although they show sinus rhythm during the time of recording. In surface ECG such markers have been suspected. The use of esophageal long-term electrocardiography with its better signal properties is a promising alternative to find such surrogate markers for risk stratification.

Objective

Identification and characterization of surrogate markers indicative for pAF in patients with sinus rhythm at the time of recording.

Methods

A total of 60 patients will be included to identify and characterize surrogate markers for pAF. Cases with known pAF will consecutively be recruited from the cardiology ward and the cardiological ambulatory. After inclusion, an age (+/- one year) and gender adjusted control person without known pAF (negative 7-day ECG within the previous 365 days before study inclusion) will be matched to every patient. Cases and controls will receive a simultaneous 24-hour esophageal electrocardiography and standard surface electrocardiography. Controls without negative 7-day ECG within the past year will have to wear the surface ECG recorder for additional 6 days (total surface ECG recording of 7 days). In the case that paroxysmal atrial fibrillation is detected for the very first time during the study, patients will be allocated to the "case" group.

Additionally, in all patients LA diameter parasternal will be measured echocardiographically.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Written informed consent
* Hospitalized patient on the cardiology ward or referred to the cardiological ambulatory
* Paroxysmal atrial fibrillation but in sinus rhythm at the time of inclusion (cases)
* Sinus rhythm without known heart rhythm disorders (controls)

Exclusion Criteria

* Persistent atrial fibrillation
* Pacemaker/ICD with atrial electrode
* History of ablation of atrial fibrillation
* Instable angina pectoris/acute myocardial infarction before revascularisation
* Cardiorespiratory unstable patients
* History of heart transplantation
* Known severe bleeding diathesis
* Carcinoma of the esophagus or nasopharynx
* Pregnancy
* History of valve replacement operation less than 4 weeks ago
* Obstructive cardiomyopathy with severe dynamic LVOT-obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients hospitalized on the cardiology ward (for any reasons). Additionally, also patients referred to the cardiology ambulatorium for a long-term ECG will be asked to participate the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number atrial premature beats not conducted to the ventricles | during analysis of the ECG

SECONDARY OUTCOMES:
Mean duration of the p-eso-wave | during analysis of the esophageal ECG
Mean duration of the left atrial wavefront | during analysis of the esophageal ECG
p-eso-wave-duration-dispersion | during analysis of the esophageal ECG
mean number of p-eso-wave-peaks | during analysis of the esophageal ECG
root mean square voltages of the last 20 ms of the p-eso-wave in the esophageal ECG | during analysis of the esophageal ECG

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Vogel, MD, PhD, Principal Investigator — Bern University Hospital; Andreas D Haeberlin, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Haeberlin A, Niederhauser T, Tanner H, Vogel R. Atrial waveform analysis using esophageal long-term electrocardiography reveals atrial ectopic activity. Clin Res Cardiol. 2012 Nov;101(11):941-2. doi: 10.1007/s00392-012-0477-6. Epub 2012 May 22. No abstract available. PMID 22614730